CLINICAL TRIAL: NCT06578650
Title: A Prospective, Single-arm, Clinical Trial of Electrospun Fiber Matrix (Restrata) in the Treatment of Surgical Defects Secondary to Resection of Malignant Cutaneous Neoplasms
Status: Recruiting | Type: Observational
Sponsor: Acera Surgical, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 24-RES-002
Record Dates: First submitted 2024-08-26; First posted 2024-08-29 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Surgical Wound
MeSH Terms: conditions — Surgical Wound

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Device: Synthetic Electrospun Fiber Matrix — Patients who are eligible for enrollment will be treated with Synthetic Electrospun Fiber Matrix immediately after surgical resection to the resulting wound

SUMMARY:
The goal of this observational prospective study is to evaluate wound healing outcomes in resection wounds resulting from surgical removal of cutaneous malignancies treated with a synthetic electrospun fiber matrix. This study intends to quantify the time from initial resection and product application to time of complete granulation of the wound bed in weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is at least 18 years old
2. Patient plans to undergo surgical resection of a cutaneous neoplasm
3. Patient is willing and capable of complying with all protocol requirements
4. Patient or legally authorized representative (LAR) is willing to provide written informed consent prior to participation in study
5. Post-resection surgical wound with a surface area of ≥4 cm2 and ≤ 36cm2

Exclusion Criteria:

1. Inability to give informed consent or to complete the procedures required for study completion
2. Patient has been previously enrolled into this study, or is currently participating in another drug or device study that has not reached its primary endpoint
3. Patient is pregnant, breast feeding or planning to become pregnant
4. Patient has a known allergy to resorbable suture materials, e.g. Polyglactin 910 (PGLA), Polydioxanone (PDS)
5. Patients receiving any immunotherapy, radiation, or chemotherapy within the past four weeks prior to resection surgery.
6. Patient has a life expectancy less than six months as assessed by the investigator
7. Patient has an additional non-study related wound within 3 cm of the study wound
8. Study wound is located on the hands or feet
9. Patient has been diagnosed with osteomalacia
10. Resection defect from a squamous cell carcinoma arising from a chronic wound
11. Patient has an uncontrolled thyroid disorder
12. Hgb A1c > 12% within 3 months prior to enrollment in patients with a known history of diabetes
13. Patient has a BMI > 34.9
14. Patient has used any tobacco product within the past 30 days prior to surgery
15. Patients with chronic kidney disease on peritoneal or hemodialysis, or with an estimated glomerular filtration rate less than 15mL/min
16. Patients with severe liver disease with active cirrhosis defined as a gross ascites upon clinical exam or a Model for End-stage Liver Disease (MELD)-Na score greater than 15
17. Patient not in reasonable metabolic control in the judgement of the investigator
18. Patient has a known history of poor compliance with medical treatment
19. Patient has a history of radiotherapy to wound bed of interest
20. Patient has been diagnosed with at least one of the following autoimmune connective tissue diseases: lupus, vasculitis, sickle cell, or uncontrolled rheumatoid arthritis
21. Active infection, undrained abscess, or critical colonization of the wound with bacteria in the judgement of the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be enrolled in a University Hospital Setting
Sampling Method: Non-Probability Sample
Enrollment: 34 (Estimated)
Dates: Start 2024-10-31 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Time to wound bed granulation | Weekly assessments until granulation achieved or up to 6 weeks following resection surgery
  Time from initial resection and product placement to the time of at least 75% wound bed granulation using a modified Bates-Jenson Scale. The Bates-Jenson Scale for Granulation Tissue ranges from: 1=Skin intact or partial thickness wound, to: 5=No granulation tissue present. Wounds are considered "granulated" upon receiving a rating of 2 (Bright, beefy red;75% to 100% of wound filled &/or tissue overgrowth) or less upon investigator assessment. Lower scores are indicative of better outcomes.

SECONDARY OUTCOMES:
Time to complete wound healing | Until healed or until 16 weeks post resection
  Total healing time will be documented (in days) at the final follow-up appointment by calculating the difference using the resection visit and "healed" visit dates.
Patient pain | Weekly for up to six weeks post resection
  Pain reported by patient on a Visual Analogue Scale (VAS), with 0 indicating no pain and 10 indicating worst pain possible. Lower scores are indicative of a better outcome
Time to skin grafting | Weekly for up to 6 weeks post-resection
  Time from resection and product place until skin grafting (if patient elects to do so)
Skin graft "take" rate | 1 week after skin graft application
  Percent of skin graft incorporation as assessed by the investigator, in patients who elect to undergo skin grafting
Tissue flap take rate | 1 week after tissue flap procedure
  Percent of successful tissue graft incorporation as assessed by the investigator, in patients who elect to undergo tissue flap procedures

OTHER OUTCOMES:
Scar quality | At the time of complete wound closure and at the 6 month post-resection follow up
  Scar quality using a Vancouver Scar Scale (VSS). The scale ranges from 0 (normal skin) to 13 (worst scar outcome). Lower scores are indicative of a better scar outcome
Infection rate and severity | to be assessed at each visit for up to 6 months post resection
  Incidence and severity of wound bed infection (if one occurs) per CTCAE V5.0 definitions ranging from 1 (localized, local intervention indicated) to 5 (death). Lower scores are indicative of milder infections
Skin Graft Failure | To be assessed at each post skin graft visit for up to 6 months post-resection
  Incidence of inadequate skin graft adherence to the underlying wound bed as assessed by the investigator in patients who have received a skin graft
Tissue flap failure | Each post-flap follow up visit for up to 6 months post-resection
  Incidence of complete flap necrosis or need for total flap removal in patients who receive a tissue flap
Incidence of local skin cancer recurrence | at the 6 month post-resection follow up
  local recurrence of skin cancer

CONTACTS AND LOCATIONS:
Locations (1):
- University Nevada - Las Vegas, Las Vegas, Nevada, United States

IPD SHARING:
Plan to Share IPD: No